CLINICAL TRIAL: NCT02615665
Title: Role of CD3+ and NKp46+ Cells in Resected Colorectal Liver Metastases.
Brief Title: Intratumoral CD3+ and NKp46+ Cells in Colorectal Liver Metastases
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Professor of Surgery, University of Milan
Other Study IDs: NKTCellsInCLM
Record Dates: First submitted 2015-11-18; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Liver Metastases
Keywords: NK-cells; T-cells
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — We use the surgical specimens.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Hepatic resection — Removal of a part of the liver during surgery
  Other Names: Hepatectomy; liver resection; liver surgery

SUMMARY:
The long-term outcome of patients resected for colorectal liver metastases (CLM) after neoadjuvant chemotherapy (CHT) depends by several tumoral and non-tumoral factors, such as the immune response to the tumor and to the CHT. The aim of this study was to investigate the impact of the pathological and immunological response in patients undergoing liver resection for CLM after CHT in regards to the long-term outcome.

DETAILED DESCRIPTION:
The immunoreactivity to CD3+ and NKp46+ cells inside the tumor, at the border between the tumor and the normal liver, and inside the normal liver will be tested by computer-assisted image analyses in patients undergoing liver resection for CLM between 2005 and 2013 preoperatively treated with oxaliplatin or irinotecan with or without bevacizumab or cetuximab. The survival will be assessed in relation to several prognostic factors and to that immunoreactivity.

ELIGIBILITY:
Inclusion Criteria:

* histological proven colorectal liver metastases
* complete clinical, surgical, pathological and follow-up data

Exclusion Criteria:

* non-radical surgery
* incomplete clinical, surgical, pathological and follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal liver metastases scheduled for surgery at our Unit.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD, PhD, Principal Investigator — Humanitas University, Humanitas Research Hospital IRCCS
Locations (1):
- Department of Hepatobiliary and General Surgery, Humanitas Research Hospital, University of Milan, Rozzano, Milan, Italy

REFERENCES:
- [Result] Hudspeth K, Donadon M, Cimino M, Pontarini E, Tentorio P, Preti M, Hong M, Bertoletti A, Bicciato S, Invernizzi P, Lugli E, Torzilli G, Gershwin ME, Mavilio D. Human liver-resident CD56(bright)/CD16(neg) NK cells are retained within hepatic sinusoids via the engagement of CCR5 and CXCR6 pathways. J Autoimmun. 2016 Jan;66:40-50. doi: 10.1016/j.jaut.2015.08.011. Epub 2015 Aug 30. PMID 26330348
- [Result] Hudspeth K, Pontarini E, Tentorio P, Cimino M, Donadon M, Torzilli G, Lugli E, Della Bella S, Gershwin ME, Mavilio D. The role of natural killer cells in autoimmune liver disease: a comprehensive review. J Autoimmun. 2013 Oct;46:55-65. doi: 10.1016/j.jaut.2013.07.003. Epub 2013 Jul 21. PMID 23880068